CLINICAL TRIAL: NCT05416723
Title: Occupational and Environmental Origins of ANCA Vasculitis: Contribution of Data From the National Network for Vigilance and Prevention of Occupational Pathologies (RNV3P)
Acronym: ANCAPRO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ANCAPRO (29BRC22.0035)
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-04

CONDITIONS: ANCA Associated Vasculitis; Occupational Diseases; Environmental Exposure
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Occupational Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to identify specific risk factors for ANCA vasculitis of occupational and/or environmental origin (exposures identified by questioning, geographical distribution of cases) from the RNV3P data.

The secondary objectives are as follows:

* Description of cases of ANCA vasculitis seen in French occupational pathology consultation centres:

  * reasons for consultation,
  * occupational and environmental etiologies described
  * occupational situations responsible
  * aptitude notices
  * recognition as an occupational disease
* Identification of specific risk factors for ANCA vasculitis of occupational and/or environmental origin (exposures identified on questioning, geographical distribution of cases).
* For occupational and non-occupational cases of ANCA vasculitis: identification of difficulties encountered by patients at work and proposed work adaptations.
* Estimation of the number of applications for recognition of disabled worker status made within this patient group.
* Identification of clinical severity and autoimmune profiles of ANCA vasculitis of occupational and/or environmental origin.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ANCA vasculitis defined according to the International Classification of Diseases (ICD-10), i.e. M 308, M 31, N 057 and L 95, or mentioned as the reason for consultation in the text mining summary.
* Seen in consultation in the occupational disease consultation centres belonging to the RNV3P
* No opposition

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ANCA vasculitis seen in French occupational disease consultation centres.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of diagnoses of ANCA vasculitis in the RNV3P | 4 months
  Number of diagnoses of ANCA vasculitis coded in the RNV3P or mentioned as the disease motivating the consultation in the summary by text mining search.

SECONDARY OUTCOMES:
Imputability of the coded diagnoses of ANCA vasculitis. | 4 months
  Number of patients with ANCA vasculitis seen in consultation in occupational disease consultation centres for which a link between occupational and/or environmental exposure and the patient's ANCA vasculitis was retained. The imputability is coded in the RNV3P database by the clinician who saw the patient, for each exposure recorded in the database, according to the pathology selected and the patient's exposure following the completion of the patient's laboris and environmental curriculum.
Number of patients with ANCA vasculitis for whom occupational and/or environmental exposure to microcrystalline silica was identified. | 4 months
  Number of patients with ANCA vasculitis seen in consultation in occupational disease consultation centres for whom occupational and/or environmental exposure to microcrystalline silica was identified.
Number of patients with ANCA vasculitis for whom other occupational and/or environmental exposure was identified. | 4 months
  Number of patients with ANCA vasculitis seen in consultation in occupational disease consultation centres for whom other occupational and/or environmental exposure was identified.
Number of patients with ANCA vasculitis for whom an application for recognition as a disabled worker has been submitted. | 4 months
  Number of patients with ANCA vasculitis seen in consultation in occupational disease consultation centres for whom an application for recognition as a disabled worker has been submitted.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU de Bordeaux, Bordeaux
  - CHU de Grenoble, Grenoble
  - CHU de LILLE, Lille
  - HCL, Lyon
  - AP-HM, Marseille
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Cochin ( AP-HP), Paris
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 3 months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.